CLINICAL TRIAL: NCT01471925
Title: A Phase III, Randomized, Open-label, Superiority Study Comparing the Incremental Product Esomeprazole Associated With Sodium Bicarbonate Made by Eurofarma and Nexium® in the Treatment of Gastroesophageal Reflux Disease
Brief Title: Study Comparing Esomeprazole Associated With Sodium Bicarbonate From Eurofarma and Esomeprazole in Treatment of Gastroesophageal Reflux Disease ESOBIC
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Change company strategy
Sponsor: Eurofarma Laboratorios S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EF 095
Record Dates: First submitted 2011-10-31; First posted 2011-11-16 (Estimated); Last update posted 2025-04-01 (Actual); Status verified 2011-11

CONDITIONS: Gastroesophageal Reflux Disease
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — Esomeprazole; Omeprazole; Sodium Bicarbonate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Esomeprazole (40mg) + Sodium Bicarbonate (721mg) (Experimental)
  Interventions: Drug: Esomeprazol (40mg) + Sodium Bicarbonate (721mg)
- Nexium® (Active Comparator)
  Interventions: Drug: Nexium®

INTERVENTIONS:
Drug: Nexium® — The medication, esomeprazole magnesium trihydrate (40 mg), should be administered once a day (before breakfast) and the capsules should be taken on an empty stomach (orally) with liquid (water at room temperature - 200 to 250 ml.
  The study treatment will last a total of 28 days.
  Arms: Nexium®
Drug: Esomeprazol (40mg) + Sodium Bicarbonate (721mg) — The medication, Esomeprazol (40 mg) + Sdium Bicarbonate (721 mg), should be administered once a day (before breakfast) and the capsules should be taken on an empty stomach (orally) with liquid (water at room temperature - 200 to 250 ml.
  The study treatment will last a total of 28 days.
  Arms: Esomeprazole (40mg) + Sodium Bicarbonate (721mg)

SUMMARY:
A phase III, randomized, open-label, superiority study comparing the incremental product esomeprazole associated with sodium bicarbonate made by Eurofarma and Nexium® in the treatment of gastroesophageal reflux disease. The study will enroll 94 patients in each arm (total of 188 patients).

ELIGIBILITY:
Inclusion Criteria:

ICF signing;

* Age ≥ 18 years;
* Gastroesophageal reflux disease diagnosis;
* Grade 0 to grade III reflux esophagitis, assessed by means of upper gastrointestinal endoscopy;
* Ability to have the endoscopy, pH-metry and esophageal manometry examinations performed;
* Washout period of 1 week without using PPI, H2 antagonists and prokinetic agents and of at least 1 day without using antacids.

Exclusion Criteria:

* Presence of esophagitis requiring intervention (grade IV), esophageal varices, Barrett's esophagus, systemic sclerosis or ulcers (gastric or duodenal ulcers);
* Previous gastric or esophageal surgery;
* Dietary sodium restriction, metabolic alkalosis, hypokalemia, Barter syndrome; Pregnancy or breastfeeding;
* Concomitant diseases, such as kidney, liver and heart failure;
* Suspected or confirmed cancer of any type;
* Abusive drug or alcohol use;
* Abnormal values for white blood cells, platelets or hemoglobin;
* Significant changes in serum sodium, potassium, calcium or creatinine concentrations;
* Treatment with PPI, H2 antagonists or prokinetic agents that may not be withheld during the washout period of 1 week or during the study;
* Intolerance or allergy to any of the components in the drug products assessed in the study;
* Use of nonsteroidal anti-inflammatory drugs (NSAIDs), antiemetic agents, macrolide antibiotics and systemic corticoids for a period equal to or greater than 2 weeks before the study or that is expected to require prolonged use during study treatment;
* Concomitant use or requirement of a gastric pH-dependent medication for optimal absorption;
* Scheduled use of other medications metabolized by cytochrome CYP during the study;
* History of active peptic ulcer;
* Rare hereditary problems of fructose intolerance, glucose-galactose malabsorption or sucrose-isomaltase insufficiency;
* Recent participation (within the last 12 months) in another clinical study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
Efficacy | 1 month
  Primary efficacy analysis the value for intragastric pH 10 centimeters distant from the lower esophageal sphincter and the pH value 1 hour after using study medication during randomization visit will be considered for primary study assessment.

CONTACTS AND LOCATIONS:
Locations (6):
- Brazil (6):
  - Instituto Goiano de Gastroenterologia, Goiânia, Goiás
  - Centro de pesquisa Clínica do Serviço de gastroenterologia, Rio de Janeiro, Rio de Janeiro
  - Mãe de Deus Center, Porto Alegre, Rio Grande do Sul
  - Centro de Pesquisa Clínica de Campinas, Canpinas, São Paulo
  - Centro de Estudos Clínicos do Interior Paulista, Jaú, São Paulo
  - Hospital Israelita Albert Einstein, São Paulo, São Paulo